CLINICAL TRIAL: NCT06996769
Title: Constrain Induced Therapy to Improve Motor Function and Body Balance in Patients With Stroke
Brief Title: Constraint-Induced Movement Therapy After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanan Hosny M Battesha (Other)
Responsible Party: Sponsor-Investigator, Hanan Hosny M Battesha, associate professor hanan hosny M Battesha, Al-Zaytoonah University of Jordan
Organization: Al-Zaytoonah University of Jordan (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STROKE
Record Dates: First submitted 2025-05-04; First posted 2025-05-30 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Hemiplegia Following Ischemic Stroke
Keywords: Constraint-Induced Movement; stroke; motor function; body balance
MeSH Terms: conditions — Stroke | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator)
  Interventions: Other: Conventional therapy for stroke patient
- intervention (Experimental): intervenstion study
  Interventions: Other: constraint induced therapy

INTERVENTIONS:
Other: constraint induced therapy — Constraint induced movement therapy (CIMT) is a treatment approach that can be used with patients who have had a CVA. In order to be eligible for the therapy, the clients must have at least 10 degrees of active wrist and finger extension. During this treatment the unaffected limb is restrained (usually with a sling or a mitt) for 90% of their waking hours. This treatment forces the client to use the affected limb throughout their daily tasks in order to combat learned non-use of the affected limb.
  Arms: intervention
Other: Conventional therapy for stroke patient — general exercises
  Arms: control group

SUMMARY:
Constraint-induced movement therapy (CIMT) is a neurological rehabilitation treatment designed to improve upper and lower extremities motor functions after stroke. The basis of CIMT is improving the function of the affected limb after a stroke by restricting the use of the healthy limb and forcing the use of the affected side. The core strategy of CIMT is the application of movement techniques, behavioral techniques and restriction methods to increase the frequency of use of the affected limb in stroke patients, improve the quality of movement of the affected limb in real-life scenarios, prevent or correct the learned non-use of the affected limb, and promote the recovery of motor function in the affected limb. This method induces the use of the affected limb, corrects or reverses habitual disuse and neglect of the affected limb, and provides structural and functional training and repeated practice opportunities for the affected limb.

ELIGIBILITY:
Inclusion Criteria:

* grade 1 or 1+ modified ashower scale
* Walk independently

Exclusion Criteria:

* moderate to sever spasticity
* balance dysfunction

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
motor function | 4 weeks
  scale to measure activity of daily lining of upper limb and lower limb and trunk control; when the number of scores increases, that means patient better

CONTACTS AND LOCATIONS:
Locations (1):
- Al Zaytoonah University, Amman, Jordan